CLINICAL TRIAL: NCT03761797
Title: Post Marketing Surveillance in Japan on Long Term Drug Use of TRADIANCE® Combination Tablets AP and BP in Patients With Type 2 Diabetes Mellitus
Brief Title: A Long-term Study on the Side Effects of TRADIANCE in Japanese Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 1275-0026
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Results first posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with type 2 Diabetes Mellitus
  Interventions: Drug: TRADIANCE® Combination Tablets AP; Drug: TRADIANCE® Combination Tablets BP

INTERVENTIONS:
Drug: TRADIANCE® Combination Tablets AP — Fixed dose combination
Drug: TRADIANCE® Combination Tablets BP — Fixed dose combination

SUMMARY:
Study objectives is to investigate the safety of long-term daily use of TRADIANCE® Combination Tablets AP and BP in Japanese patients with Type 2 Diabetes mellitus (T2DM) used in routine care.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients with Type 2 Diabetes mellitus (T2DM) who are prescribed with TRADIANCE® Combination Tablets AP or BP
* Patients who have never been treated with TRADIANCE® Combination Tablets AP or BP before enrolment

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 2 Diabetes Mellitus
Sampling Method: Non-Probability Sample
Enrollment: 1164 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rie Ikeda, 81364172200, Study Chair — zzCDMJP_PV_PMS@boehringer-ingelheim.com
Locations (1):
- Nippon Boehringer Ingelheim Co., Ltd, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https:// trials.boehringer-ingelheim.com/trial_results/ clinical_submission_documents.html to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Also, Researchers can use the following link http://trials.boehringeringelheim. com/ to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website. The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Inagaki N, Nishimoto T, Nishiya Y, Nitta D. Safety and effectiveness of empagliflozin and linagliptin fixed-dose combination therapy in Japanese patients with type 2 diabetes: final results of a one-year post-marketing surveillance study. Expert Opin Drug Saf. 2023 Feb;22(2):153-163. doi: 10.1080/14740338.2022.2107200. Epub 2022 Aug 16. PMID 35946927
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-interventional study based on newly collect data of patients under routine care to confirm safety of TRADIANCE® Combination Tablets AP and BP in real-world setting in Japanese patients with Type 2 Diabetes mellitus (T2DM).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- All Patients With Type 2 Diabetes Mellitus: TRADIANCE® Combination Tablet AP or BP (fixed dose combination of empagliflozin and linagliptin) were administered orally once daily for patients with type 2 Diabetes Mellitus (T2DM). The TRADIANCE® Combination Tablet AP contains 10 milligrams (mg) empagliflozin and 5 mg linagliptin, while Tablet BP contains 25 mg empagliflozin and 5 mg linagliptin. Patients were followed up to 52 weeks.
Period: Overall Study
Arm/Group | All Patients With Type 2 Diabetes Mellitus
Started | 1164
Safety Set | 1146
Completed | 1025
Not Completed | 139
Not completed — Changing hospital | 11
Not completed — Improvement/remission | 6
Not completed — Withdrawal by Subject | 19
Not completed — Lost to Follow-up | 33
Not completed — Adverse Event | 37
Not completed — Case report form (CRF) not collected | 5
Not completed — No patient visit after entry | 13
Not completed — Switch to other diabetes medication | 10
Not completed — Prevention for recurrence of cystitis | 1
Not completed — Postoperative therapy of esophageal cancer | 1
Not completed — Insufficient effectives | 2
Not completed — Excessive alcohol intake | 1

BASELINE CHARACTERISTICS:
Population: Safety set: The safety set included all patients who had no invalid registration, who were documented to have taken at least one dose of TRADIANCE® Combination Tablets AP or BP.
Arm/Group | All Patients With Type 2 Diabetes Mellitus
Number analyzed (Participants) | 1146
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.8 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 394
  Male | 752
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reactions (ADRs)
Description: The number of participants with adverse drug reactions is reported.
Time Frame: From first dose of study medication until last dose + 7 days, up to 102.1 weeks.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients With Type 2 Diabetes Mellitus
Number analyzed (Participants) | 1146
Participants | 32

ADVERSE EVENTS:
Time Frame: From first dose of study medication until last dose + 7 days, up to 102.1 weeks.
Description: Safety set: The safety set included all patients who had no invalid registration, who were documented to have taken at least one dose of TRADIANCE® Combination Tablets AP or BP.
Arm/Group | All Patients With Type 2 Diabetes Mellitus
All-Cause Mortality (participants affected / at risk) | 5/1146
Serious Adverse Events (participants affected / at risk) | 40/1146
Other Adverse Events (participants affected / at risk) | 0/1146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients With Type 2 Diabetes Mellitus (N=1146)
Infective spondylitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Pyoderma (Infections and infestations) | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Carotid artery occlusion (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Atrioventricular block second degree (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Idiopathic interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Cholangitis acute (Hepatobiliary disorders) | 1
Death (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Pneumonia bacterial (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Cerebral infarction (Nervous system disorders) | 4
Thalamic infarction (Nervous system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Myocarditis (Cardiac disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Parathyroid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Scrotal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT03761797/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT03761797/SAP_001.pdf